CLINICAL TRIAL: NCT00886899
Title: Facilitated Antegrade Steering Technique in Chronic Total Occlusions
Brief Title: Facilitated Antegrade Steering Technique in Chronic Total Occlusions (FAST-CTOs)
Acronym: FAST-CTOs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BridgePoint Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200-0002
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Chronic Total Occlusion
Keywords: CTO; chronic total occlusion; CAD; coronary artery disease; interventional cardiology; revascularization; recanalization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BridgePoint Medical System (Experimental): Attempt to cross CTO with the BridgePoint Medical System after an attempt to cross the CTO with a currently marketed guidewire
  Interventions: Device: Recanalization of a coronary chronic total occlusion

INTERVENTIONS:
Device: Recanalization of a coronary chronic total occlusion — Crossing a CTO to allow definitive treatment via balloon angioplasty and/or stent placement
  Other Names: CrossBoss Catheter; Stingray Catheter; Stingray Guidewire

SUMMARY:
Prospective, non-randomized, multicenter study in subjects with coronary artery chronic total occlusions (CTOs). Published results of safety and effectiveness of conventional techniques will be used for comparison. Enrollment of up to 149 subjects with a CTO refractory to currently marketed guidewire use and meeting all inclusion/exclusion criteria at up to 15 US clinical sites. Hypothesis is that the BridgePoint Medical System is safe and effective in treating coronary CTOs compared to CTO literature.

ELIGIBILITY:
Inclusion Criteria:

* suitable candidate for non-emergent, coronary angioplasty
* documented coronary CTO lesion with the following characteristics: a) Thrombolysis in Myocardial Infarction (TIMI) 0 flow for at least 90 days; b) satisfactory distal vessel visualization; and c) refractory to currently marketed guidewire crossing via 1 of the following: 1. previous failed attempt to cross CTO within the past 12 months; or 2. unsuccessful CTO crossing w/ guidewire (10-15 min fluoro time); or 3. attempt to cross CTO w/ guidewire results in subintimal guidewire
* angina or ischemia caused by the occluded artery
* at least 18 years of age
* Body Mass Index (BMI) < 40
* left ventricle ejection fraction > 20%
* sign the Informed Consent Form

Exclusion Criteria:

* saphenous vein graft (SVG) CTO or an in-stent CTO
* aorto-ostial CTO location. (Ostial bifurcation origins may be considered)
* intolerance to aspirin or a neutropenic response to Ticlopidine/Clopidogrel
* appearance of thrombus or intraluminal filling defects
* severe cerebrovascular disease (history of stroke or TIA within 1 month)
* cardiac intervention within two weeks of the procedure
* renal insufficiency (serum creatinine of > 2.3 mg/dl)
* active gastrointestinal bleeding
* active infection or fever that may be due to infection
* life expectancy < 2 years due to other illnesses
* significant anemia (hemoglobin < 8.0 mg / dl)
* severe uncontrolled systemic hypertension
* severe electrolyte imbalance
* anaphylaxis to angiographic contrast media unless appropriately medicated
* congestive heart failure [New York Heart Association (NYHA) Class IV]
* unstable angina requiring emergent percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG)
* recent myocardial infarction (MI)(within the past two weeks)
* uncontrolled diabetes
* participation in another investigational protocol
* unwillingness or inability to comply with any protocol requirements
* pregnant or nursing
* extensive dissection from refractory guidewire use
* crossing CTO (true lumen) w/ guidewire within 10-15 min of fluoro time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Whitlow, MD, Principal Investigator — The Cleveland Clinic
Locations (16):
- United States (16):
  - St. Luke's Medical Center, Phoenix, Arizona
  - Scripps Clinic, La Jolla, California
  - University of California Davis Heart & Vascular Center, Sacramento, California
  - Stanford University Hospital, Stanford, California
  - Torrance Memorial Medical Center, Torrance, California
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Prairie Cardiovascular Consultants, Springfield, Illinois
  - Minneapolis Heart Institute, Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic - St. Mary's Hospital, Rochester, Minnesota
  - Mid America Heart Institute, St. Luke's Hospital, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Dallas VA Medical Center, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - St. Joseph Hospital, Bellingham, Washington

REFERENCES:
- [Derived] Whitlow PL, Burke MN, Lombardi WL, Wyman RM, Moses JW, Brilakis ES, Heuser RR, Rihal CS, Lansky AJ, Thompson CA; FAST-CTOs Trial Investigators. Use of a novel crossing and re-entry system in coronary chronic total occlusions that have failed standard crossing techniques: results of the FAST-CTOs (Facilitated Antegrade Steering Technique in Chronic Total Occlusions) trial. JACC Cardiovasc Interv. 2012 Apr;5(4):393-401. doi: 10.1016/j.jcin.2012.01.014. PMID 22516395

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BridgePoint Medical System
Started | 147
Completed | 147
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BridgePoint Medical System
Number analyzed (Participants) | 147
Age Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 127
Region of Enrollment [Number; unit: participants]
  United States | 147

OUTCOME MEASURES:

1. Primary Outcome: Technical Success
Description: Defined as the ability of the BridgePoint Medical System to successfully facilitate placement of a guidewire beyond a chronic total occlusion (CTO) in the true vessel lumen in cases that were otherwise refractory to treatment with a currently marketed guidewire
Time Frame: Intraprocedural
Population: Three participants had two CTOs, so there were a total of 150 CTOs in 147 participants.
Measure: Number (90% Confidence Interval); unit: percentage of CTOs
Units Other Than Participants: CTOs
Arm/Group | BridgePoint Medical System
Number analyzed (Participants) | 147
Number analyzed (CTOs) | 150
percentage of CTOs | 77 [70 to 82]

2. Primary Outcome: 30-day Major Adverse Cardiac Event (MACE) Rate
Description: Defined as cardiac death, Q-wave and non-Q-wave [total creatinine kinase (CK) >2x upper limit of normal with a positive myocardial band (MB) fraction] myocardial infarction (MI), target lesion revascularization (TLR), and emergency bypass surgery.
Time Frame: 30 Days
Population: Includes 21 patients with "early" (<30 day) follow-up
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | BridgePoint Medical System
Number analyzed (Participants) | 147
percentage of participants
  All participants | 4.8 [2.3 to 8.8]
  Patients with at least 30-days follow-up (n=136) | 5.1 [2.5 to 9.5]

3. Secondary Outcome: Total Procedure Time
Description: Minus any time to determine CTO was refractory to standard guidewire
Time Frame: Intraprocedural
Population: Procedure time data for two participants was not available.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BridgePoint Medical System
Number analyzed (Participants) | 145
minutes | 105 (54)

4. Secondary Outcome: Total Procedural Fluoroscopy Time
Description: Minus any time to determine CTO was refractory to standard guidewire
Time Frame: Intraprocedural
Population: Fluoroscopy time was not available for two participants
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BridgePoint Medical System
Number analyzed (Participants) | 145
minutes | 44 (25)

ADVERSE EVENTS:
Arm/Group | BridgePoint Medical System
Serious Adverse Events (participants affected / at risk) | 25/147
Other Adverse Events (participants affected / at risk) | 61/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BridgePoint Medical System (N=147)
Death (Cardiac disorders) | 2 (2)
Non-Q-Wave Myocardial Infarction (NQWMI) (Cardiac disorders) | 6 (6) — Defined as total serum creatinine kinase (CK) greater than twice the upper limit of normal with greater than the upper limit of normal myocardial band (CK-MB)
Cerebral Vascular Accident/Stroke (Nervous system disorders) | 1 (1)
Perforation (Vascular disorders) | 10 (10)
Pericardial Effusion (Cardiac disorders) | 3 (3)
Arrhythmia Requiring Treatment (Cardiac disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BridgePoint Medical System (N=147)
Cardiac Enzyme Elevation (Cardiac disorders) | 21 (21) — Enzyme elevation that did not fit the definition of NQWMI
Untreated Dissection (Vascular disorders) | 1 (1)
Puncture Site Complication (Vascular disorders) | 11 (11)
Non-Target Vessel Treatment (Vascular disorders) | 3 (3)
Other (Vascular disorders) | 25 (25) — Includes but not limited to: chest pain, hypotension, radiation burn, pulmonary embolism, dermatitis, vomiting, vasovagal reaction, and heart murmur.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No